CLINICAL TRIAL: NCT03736174
Title: The Utilization of High Frequency Ultrasound to Diagnose Chronic Exertional Compartment Syndrome: A Pilot Study
Brief Title: Utilization of High Frequency Ultrasound to Diagnose Chronic Exertional Compartment Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-1297
Record Dates: First submitted 2018-10-30; First posted 2018-11-09 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Chronic Exertional Compartment Syndrome
Keywords: CECS
MeSH Terms: conditions — Chronic Exertional Compartment Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Compartment Pressure Testing: Patients who present with symptoms of CECS will be consented and tested per protocol with compartment pressure testing. Concurrently, patients will undergo a high frequency ultrasound to observe any patterns in structure to assist future research in noninvasively diagnosing CECS. Evaluation of ultrasonographic findings will be dependent on tissue density as measured by hypoechoic versus hyperechoic signal as well as muscle compartment thickness at its largest dimension.
- Control: Control subjects will undergo exercise protocol and ultrasound, but will not have compartment pressure testing completed.

SUMMARY:
The purpose of this study is to investigate high frequency ultrasound as a future modality for the diagnosis of chronic exertional compartment syndrome (CECS). The results of the ultrasound will help determine if there are any significant radiologic findings or patterns seen in patients with CECS.

DETAILED DESCRIPTION:
The purpose of this study is to investigate high frequency ultrasound as a future modality for the diagnosis of chronic exertional compartment syndrome (CECS). The results of the ultrasound will help determine if there are any significant radiologic findings or patterns seen in patients with CECS. Evaluation of ultrasonographic findings will be dependent on tissue density as measured by hypoechoic versus hyperechoic signal as well as muscle compartment thickness at its largest dimension. A specific aim for this study would be to facilitate future research in order to eliminate the need for painful and invasive diagnostic techniques for CECS.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 13 and over
* Patients with any combination of the following symptoms who would otherwise be evaluated for CECS:
* Symptoms of leg pain worsened with activity and relieved by rest
* Pain that is generalized in the anterior or lateral compartments of lower leg
* Numbness or tingling in the distribution of the superficial peroneal nerve
* Sensation of "slap foot" or anterior/lateral compartment weakness
* Able to exercise for CPT testing: Patients will be asked to go through a standardized warm up on a treadmill with increasing speed and incline settings until symptoms are achieved. They will maintain exercise for a minimum of five minutes or to patient tolerance.

Exclusion Criteria:

* Known vascular disease
* Neurogenic or radicular symptoms

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are seen at the University of Colorado Sports Medicine Clinic who present with symptoms of CECS.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-12-07 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Ultrasound to predict/diagnose CECS | 2 weeks
  Determine if there are significant radiologic patterns arising on ultrasound imaging to help further future research predict or diagnose CECS using non-invasive methods.Specific aim is to investigate high frequency ultrasound as a future modality for the diagnosis of CECS. The results of the ultrasound will help determine if there are any significant radiologic findings or patterns seen in patients with CECS

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Wolcott, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado - Sports Medicine, Denver, Colorado, United States

REFERENCES:
- [Background] Aweid O, Del Buono A, Malliaras P, Iqbal H, Morrissey D, Maffulli N, Padhiar N. Systematic review and recommendations for intracompartmental pressure monitoring in diagnosing chronic exertional compartment syndrome of the leg. Clin J Sport Med. 2012 Jul;22(4):356-70. doi: 10.1097/JSM.0b013e3182580e1d. PMID 22627653
- [Background] Barnes M. Diagnosis and management of chronic compartment syndromes: a review of the literature. Br J Sports Med. 1997 Mar;31(1):21-7. doi: 10.1136/bjsm.31.1.21. No abstract available. PMID 9132204
- [Background] Fraipont MJ, Adamson GJ. Chronic exertional compartment syndrome. J Am Acad Orthop Surg. 2003 Jul-Aug;11(4):268-76. doi: 10.5435/00124635-200307000-00006. PMID 12889865
- [Background] Gershuni DH, Gosink BB, Hargens AR, Gould RN, Forsythe JR, Mubarak SJ, Akeson WH. Ultrasound evaluation of the anterior musculofascial compartment of the leg following exercise. Clin Orthop Relat Res. 1982 Jul;(167):185-90. PMID 7094462
- [Background] Lynch JE, Heyman JS, Hargens AR. Ultrasonic device for the noninvasive diagnosis of compartment syndrome. Physiol Meas. 2004 Feb;25(1):N1-9. doi: 10.1088/0967-3334/25/1/n01. PMID 15005334
- [Background] Paik RS, Pepple DA, Hutchinson MR. Chronic exertional compartment syndrome. BMJ. 2013 Jan 15;346:f33. doi: 10.1136/bmj.f33. No abstract available. PMID 23321416
- [Background] Pedowitz RA, Hargens AR, Mubarak SJ, Gershuni DH. Modified criteria for the objective diagnosis of chronic compartment syndrome of the leg. Am J Sports Med. 1990 Jan-Feb;18(1):35-40. doi: 10.1177/036354659001800106. PMID 2301689
- [Background] Rajasekaran S, Beavis C, Aly AR, Leswick D. The utility of ultrasound in detecting anterior compartment thickness changes in chronic exertional compartment syndrome: a pilot study. Clin J Sport Med. 2013 Jul;23(4):305-11. doi: 10.1097/JSM.0b013e3182856046. PMID 23558330
- [Background] Roberts A, Franklyn-Miller A. The validity of the diagnostic criteria used in chronic exertional compartment syndrome: a systematic review. Scand J Med Sci Sports. 2012 Oct;22(5):585-95. doi: 10.1111/j.1600-0838.2011.01386.x. Epub 2011 Sep 13. PMID 22092446
- [Background] Roscoe D, Roberts AJ, Hulse D. Intramuscular compartment pressure measurement in chronic exertional compartment syndrome: new and improved diagnostic criteria. Am J Sports Med. 2015 Feb;43(2):392-8. doi: 10.1177/0363546514555970. Epub 2014 Nov 18. PMID 25406302
- [Background] Tucker AK. Chronic exertional compartment syndrome of the leg. Curr Rev Musculoskelet Med. 2010 Sep 2;3(1-4):32-7. doi: 10.1007/s12178-010-9065-4. PMID 21063498
- [Background] van den Brand JG, Nelson T, Verleisdonk EJ, van der Werken C. The diagnostic value of intracompartmental pressure measurement, magnetic resonance imaging, and near-infrared spectroscopy in chronic exertional compartment syndrome: a prospective study in 50 patients. Am J Sports Med. 2005 May;33(5):699-704. doi: 10.1177/0363546504270565. Epub 2005 Feb 16. PMID 15722275